CLINICAL TRIAL: NCT01843010
Title: Effect of Parecoxib on the Change of Shoulder Pain Threshold After Gynecological Laparoscopies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xuyu Zhang, Attending Doctor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ZSYY-2013-04-23
Record Dates: First submitted 2013-04-23; First posted 2013-04-30 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Postoperative Pain Management, Pain Threshold, Shoulder Pain, Laparoscopies
Keywords: NSAIDs; Hyperalgesia; Postlaparoscopic shoulder pain
MeSH Terms: conditions — Shoulder Pain; Hyperalgesia | interventions — parecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parecoxib (Active Comparator): Intravenously Parecoxib 40mg at 30min before intubation, 8h and 20h after surgery.
  Interventions: Drug: Parecoxib
- Placebo (Placebo Comparator): Normal saline 5ml will be intravenously infused at the same time points., respectively.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Parecoxib — Parecoxib 40mg will be intravenously infused.
  Arms: Parecoxib
Drug: Placebo — Normal saline 5ml will be intravenously infused.
  Arms: Placebo

SUMMARY:
This prospective, double blind, placebo-controlled, parallel group study will be conducted in the first affiliated hospital of Sun yat-sen university in Guangzhou, China. Patients aged 18-65 (ASA I-II) undergoing elective gynecologic laparoscopic surgery with general anesthesia will be involved in this study. According to previous studies and our pilot trial, estimated 120 patients will be involved in this study. All eligible patients will be randomly assigned to two groups. In group P, patients will receive parecoxib 40mg intravenously 30min before intubation, 8h and 20h after the surgery,respectively. In Group C, patients will receive normal saline at the same time points. The shoulder pressure pain thresholds will be measured with a pressure algometer by an independent doctor blinding to medication and grouping at the day before surgery, 24h and 48h after surgery. Moreover, the intensity of shoulder pain and side effects will be evaluated by another independent doctor at 24h and 48h after surgery. At the end of the observation, the intensity of the maximal shoulder pain will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* females age 18-65yr,
* American Society of Anesthesiologists (ASA)I-II,
* Body Mass Index(BMI) 18-25kg/m2.

Exclusion Criteria:

* a history of severe cardiac, pulmonary, hepatic, renal disease, chronic drug or alcohol abuse;
* the presence of preoperative shoulder pain or any chronic pain syndrome, long-term use of analgesics; allergy or contraindications to nonsteroidal anti-inflammatory drugs (allergy, peptic ulcer disease, gastroesophageal reflux disease, renal insufficiency, coagulopathy) and any other drugs used in the study;
* patient's pain evaluation is judged unreliable;
* patients with conversion to a laparotomy;
* refuse to coordinate with the follow-up tests.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The change of shoulder pressure pain threshold | The pressure pain thresholds are measured at the day before surgery, 24h and 48h after surgery
  The patients keep sitting position, and the pressure pain thresholds are measured twice at a fixed point in bilateral levator scapulae, supraspinatus, pectoralis major and flexor carpi ulnaris with a pressure algometer (FPX25, Wagner Instruments, USA) by an independent doctor.

SECONDARY OUTCOMES:
The severity of shoulder pain | At the day before surgery, 24h and 48h after surgery
  The patients are asked to rate the severity of shoulder pain via a visual analog scale (VAS) ranging from no pain (0) to worst possible pain (10) by another independent doctor.

CONTACTS AND LOCATIONS:
Overall Officials: Ke xuan Liu, M.D and Ph.D, Study Director — 1st affiliated hospital of Sun Yat-sen university
Locations (1):
- Department of Anesthesiology, The First Affiliated Hospital, Sun Yat-sen University., Guangzhou, Guangdong, China

REFERENCES:
- [Background] Zhang H, Shu H, Yang L, Cao M, Zhang J, Liu K, Xiao L, Zhang X. Multiple-, but not single-, dose of parecoxib reduces shoulder pain after gynecologic laparoscopy. Int J Med Sci. 2012;9(9):757-65. doi: 10.7150/ijms.4916. Epub 2012 Oct 23. PMID 23136538